CLINICAL TRIAL: NCT01912612
Title: A Study to Identify Predictors of Response to Duloxetine in Breast Cancer Patients With Chronic Pain
Brief Title: Mechanistic Study of Duloxetine in Breast Cancer Patients With Chronic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2013.044; HUM00075181 (Other: University of Michigan); HCI94979 (Other: University of Utah)
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Pain
Keywords: Breast cancer; Pain sensitivity
MeSH Terms: conditions — Pain; Breast Neoplasms | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Intervention Model Description: Trial was initially a randomized cross-over design. Soon after study initiation the trial design was amended because of poor accrual, and instead was a single arm open label trial in which all patients with pain were treated with study drug. Since so few patients had been enrolled at the time of study redesign, the only data analyzed were from the single treatment arm portion of the trial, and the non-intervention (baseline only) comparator.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Patients with pain, duloxetine) (Experimental): Duloxetine 30 mg daily x 1 week, then 60 mg daily x 4 weeks, then 30 mg daily x 2 weeks.
  Interventions: Drug: Duloxetine
- Arm 2 (Patients without pain -- control) (No Intervention): Patient reported pain and symptoms assessment for comparison at baseline.

INTERVENTIONS:
Drug: Duloxetine — Subjects will receive 30 mg duloxetine orally for 7 days, then 60 mg duloxetine orally for 28 days, then 30 mg duloxetine orally x 14 days.
  Other Names: Cymbalta
  Arms: Arm 1 (Patients with pain, duloxetine)

SUMMARY:
Early stage breast cancer is typically treated with surgery, chemotherapy, radiation therapy, and/or endocrine therapy. Following treatment, 25-60% of breast cancer survivors have reported chronic pain, which can be difficult to manage. Duloxetine is a serotonin norepinephrine reuptake inhibitor that is FDA approved for treatment of depression, anxiety, fibromyalgia, diabetic neuropathic pain, knee arthritis, and low back pain.

Pilot data suggest that duloxetine is effective in management of endocrine therapy-associated musculoskeletal pain, and a randomized placebo controlled trial of duloxetine has demonstrated efficacy for treatment of chemotherapy-induced neuropathic pain. In this mechanistic study of duloxetine, we will investigate the change in pain sensitivity with treatment in order to evaluate both why duloxetine is effective for management of pain for some patients, as well as predictors of who is likely to benefit from duloxetine. A total of 84 women with early stage breast cancer who have chronic pain following treatment, as well as 48 women who are pain free, will be enrolled. All subjects will undergo assessment of pain sensitivity and complete questionnaires. Subjects with pain will be treated with duloxetine for a total of 7 weeks, with pain sensitivity assessments before treatment and after 4 weeks of full-dose treatment.

DETAILED DESCRIPTION:
Early stage breast cancer is typically treated with surgery, chemotherapy, radiation therapy, and/or endocrine therapy. Following treatment, 25-60% of breast cancer survivors have reported chronic pain, which can be difficult to manage. Duloxetine is a serotonin norepinephrine reuptake inhibitor that is FDA approved for treatment of depression, anxiety, fibromyalgia, diabetic neuropathic pain, knee arthritis, and low back pain.

Data from a randomized, placebo-controlled clinical trial of duloxetine demonstrated that it is effective in management of both aromatase inhibitor-associated musculoskeletal pain and chemotherapy-induced neuropathic pain. In this mechanistic study, we investigated the change in pain sensitivity with treatment in order to evaluate both why duloxetine is effective for management of pain for some patients, as well as predictors of who is likely to benefit from duloxetine. The original protocol was designed as a randomized, placebo-controlled cross-over trial, with planned enrollment of a total of 84 women with early stage breast cancer who have chronic pain following treatment, as well as 48 women who are pain free. However because of challenges with logistics of the protocol and pain testing, the trial was redesigned after only 7 patients with pain were enrolled. The new design was a single arm trial, and all patients with pain were treated with duloxetine (no placebo); there was still a non-treatment comparator arm of patients without pain. Patients were enrolled first at the University of Michigan and then the University of Utah. A total of 39 patients with pain and 43 controls without pain were enrolled before the trial closed to enrollment. All subjects underwent assessment of pain sensitivity and completed questionnaires. Subjects with pain were treated with duloxetine for a total of 7 weeks, with pain sensitivity assessments before treatment and after 4 weeks of full-dose treatment. The data from the control patients (who did not receive any study medication) are being compared to those from the patients with pain to understand more about the differences between patients who do and do not experience treatment-related pain, and to interpret the post-intervention patient-reported and pain assessment results.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients at least 25 years of age
2. Diagnosis of stage 0-III breast cancer within 12 years prior to enrollment. All indicated surgery, chemotherapy, and/or radiation therapy must have been completed at least 12 weeks prior to enrollment. Concomitant endocrine therapy and targeted therapies such as palbociclib, pertuzumab, and trastuzumab are permitted.
3. Pain that developed or worsened since breast cancer diagnosis and is not due to identifiable traumatic event or fracture
4. Patient-reported worst pain score between 5 and 10 (inclusive) on a 0-10 scale (assessed verbally)
5. Female patients must be at least 1 year postmenopausal or surgically sterile; or must agree to use a medically acceptable form of contraception
6. Willing to withdraw from selective serotonin reuptake inhibitors (SSRI) and tricyclic antidepressants (TCA) prior to treatment initiation
7. Patients who are currently taking non-steroidal anti-inflammatory drugs (NSAIDs) (e.g., ibuprofen, naproxen, meloxicam, gabapentin, pregabalin) and/or opioid pain medications must remain on a stable dosage throughout the duration of the study
8. Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

1. Prior use of duloxetine or milnacipran.
2. Prior or current use of venlafaxine specifically for treatment of pain (prior or current use for treatment of other indications, such as hot flashes, is permitted, although cases currently taking venlafaxine must discontinue use prior to study treatment initiation)
3. Patients must not be taking any contraindicated medications listed on the duloxetine package insert including the following: phenothiazines, propafenone, flecainide, linezolid, or anticoagulation medication (e.g., heparin, warfarin, or direct oral anticoagulants); treatment with monoamine oxidase inhibitor within 14 days prior to registration.
4. Thumbnail abnormalities on either hand (such as due to chemotherapy or trauma, or artificial nails) that are likely to alter pain perception during testing
5. Peripheral sensory neuropathy at the thumbs bilaterally that interferes with function and/or activities of daily living
6. Significant risk of suicide based on the Investigator's judgment
7. History or behavior that would, in the Investigator's judgment, prohibit compliance for the duration of the study.
8. History of alcohol or other substance abuse or dependence within the year prior to registration
9. Known chronic liver disease, end stage renal disease, or creatinine clearance <30 mL/min as defined by Cockcroft-Gault equation
10. Uncontrolled narrow-angle glaucoma.
11. Clinically significant coagulation disorder
12. History of seizure disorder
13. Pregnant or breast-feeding. Urine pregnancy test will be assessed at the baseline visit in women of child-bearing potential with chronic pain.
14. Unable to take oral medications or any medical condition that would interfere with the absorption of study medication capsules.
15. Currently taking SSRI, serotonin-norepinephrine reuptake inhibitor (SNRI), or TCA regimen (including Wellbutrin) for treatment of major depressive disorder or generalized anxiety disorder (without approval and involvement of the patient's treating psychiatrist to taper cases off these medications prior to study treatment).

Controls are patients without chronic pain who otherwise meet the following eligibility criteria (inclusion #1, 2, 8, exclusion #1, 2, 4, 5, worst pain score 0-1, and not currently on medication for pain)

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2013-10-30 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn Henry, MD, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 3 cases randomized to placebo are not included in the analysis. See study description in protocol section for explanation. 3 patients on Arm 2 consented but withdrew prior to participation. 1 patient on Arm 1 withdrew permission to use her data.
Groups:
- Arm 1 (Patients With Pain): Duloxetine 30 mg daily x 1 week, then 60 mg daily x 4 weeks, then 30 mg daily x 2 weeks.
  Duloxetine: Subjects will receive 30 mg duloxetine orally for 7 days, then 60 mg duloxetine orally for 28 days, then 30 mg duloxetine orally x 14 days.
  Surveys administered at baseline and at 5 weeks.
- Arm 2 (Patients Without Pain -- Control): Surveys administered at baseline only.
- Arm 3 - Placebo (Withdrawn): Because of challenges with logistics of the protocol and pain testing, the trial was redesigned after only 7 patients with pain were enrolled. Three of the patients had been assigned to placebo arm. This arm is not included in any analysis.
Period: Overall Study
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control) | Arm 3 - Placebo (Withdrawn)
Started | 36 | 40 | 3
Completed | 31 | 40 | 0
Not Completed | 5 | 0 | 3
Not completed — Adverse Event | 4 | 0 | 0
Not completed — Withdrew consent | 1 | 0 | 0
Not completed — Study design change | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Population: Excluding the 1 patient in Arm 1 who withdrew consent
Groups:
- Arm 1 (Patients With Pain): Duloxetine 30 mg daily x 1 week, then 60 mg daily x 4 weeks, then 30 mg daily x 2 weeks.
  Duloxetine: Subjects will receive 30 mg duloxetine orally for 7 days, then 60 mg duloxetine orally for 28 days, then 30 mg duloxetine orally x 14 days.
- Total: Total of all reporting groups
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control) | Total
Number analyzed (Participants) | 35 | 40 | 75
Age, Continuous [Median (Full Range); unit: years] | 55 [34 to 76] | 54 [27 to 80] | 55 [27 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 40 | 75
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 35 | 40 | 75
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 2 | 2 | 4
  White | 30 | 37 | 67
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 35 | 40 | 78

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient-reported Worst Pain Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Worst pain will be assessed at baseline and 5 weeks for each individual patient using the Brief Pain Inventory.
  * Baseline: Mean worst pain for all individual patients in arm 1 (intervention) and arm 2 (control)
  * 5 weeks: Mean worst pain for all individual patients in arm 1 (intervention)
  * Range of pain score 0-10 (0=no pain; 10=worst pain)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
score on a scale
  Baseline | 6.54 (1.868) | 0.25 (0.494)
  5 weeks: number analyzed (Participants) | 31 | 0
  5 weeks | 4.06 (2.744) |

2. Secondary Outcome: Change in Patient-reported Average Pain Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Average pain will be assessed at baseline and 5 weeks for each individual patient using the Brief Pain Inventory.
  * Baseline: Mean average pain for all individual patients in arm 1 (intervention) and arm 2 (control)
  * 5 weeks: Mean average pain for all individual patients in arm 1 (intervention)
  * Range of pain score 0-10 (0=no pain; 10=worst pain)
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
score on a scale
  Baseline | 4.86 (2.088) | 0.15 (0.362)
  5 week timepoint: number analyzed (Participants) | 31 | 0
  5 week timepoint | 3.10 (2.271) |

3. Secondary Outcome: Change in Pain Interference Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Pain interference will be assessed at baseline and 5 weeks for each individual patient using the Brief Pain Inventory.
  * Baseline: Mean pain interference for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean pain interference for all individual patients in arm 1 (intervention)
  * Range of pain interference score 0-10 (0=no interference; 10=worst interference)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 had missing data at baseline and the score could not be generated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 40
score on a scale
  Baseline | 4.91 (2.09) | 0.03 (0.74)
  5 week timepoint: number analyzed (Participants) | 31 | 0
  5 week timepoint | 2.30 (2.33) |

4. Secondary Outcome: Change in Number of Sites of Pain Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Number of sites of pain will be assessed at baseline and 5 weeks for each individual patient using the Michigan Body Map.
  * Baseline: Mean number of sites of pain for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean number of sites of pain for all individual patients in arm 1 (intervention)
  * Range of number of sites of pain 0-35 (0=no pain; 35=every pre-defined body site has pain)
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Mean (Full Range); unit: number of sites
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
number of sites
  Baseline | 9.63 [1 to 22] | 0.52 [0 to 4]
  5 week timepoint: number analyzed (Participants) | 31 | 0
  5 week timepoint | 7.90 [1 to 18] |

5. Secondary Outcome: Change in Fibromyalgia Symptom Severity Score Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Fibromyalgia Symptom Severity Score will be assessed at baseline and 5 weeks for each individual patient using the Michigan Body Map and Symptom Severity Scale.
  * Baseline: Mean Fibromyalgia Symptom Severity Score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean Fibromyalgia Symptom Severity Score for all individual patients in arm 1 (intervention)
  * Range of Fibromyalgia Symptom Severity Score 0-12 (0=not consistent with fibromyalgia; 12=most consistent with fibromyalgia)
Time Frame: 5 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 40
score on a scale
  Baseline | 5.35 (2.13) | 1.68 (1.37)
  week 5 timepoint: number analyzed (Participants) | 31 | 0
  week 5 timepoint | 4.90 (2.44) |

6. Secondary Outcome: Change in PainDETECT Score Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: PainDETECT score will be assessed at baseline and 5 weeks for each individual patient using the PainDETECT questionnaire.
  * Baseline: Mean PainDETECT score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean PainDETECT score for all individual patients in arm 1 (intervention)
  * Range of PainDETECT score -1-38 (-1=no neuropathic pain; 38=most consistent with neuropathic pain)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 had missing data at baseline and 3 patients had missing data at week 5 and the scores could not be generated.
Measure: Mean (Standard Deviation); unit: score on questionnaire
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 40
score on questionnaire
  Baseline | 11.44 (8.39) | 1.13 (2.02)
  week 5 timepoint: number analyzed (Participants) | 28 | 0
  week 5 timepoint | 8.54 (8.72) |

7. Secondary Outcome: Change in Neuropathy Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Neuropathy will be assessed at baseline and 5 weeks for each individual patient using the Functional Assessment of Cancer Therapy-Gynecologic Oncology Group-Neurotoxicity (FACT/GOG-NTX) questionnaire.
  * Baseline: Mean neuropathy score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean neuropathy score for all individual patients in arm 1 (intervention)
  * Range of neuropathy score 0-44 (0=no neuropathy; 44=most consistent with neuropathy)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 at baseline, 1 patient in Arm 1 at week 5, and 1 patient in Arm 2 had missing data and the scores could not be generated.
Measure: Mean (Standard Deviation); unit: score on questionnaire
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 39
score on questionnaire
  Baseline | 14.09 (8.85) | 1.44 (1.67)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 9.10 (8.77) |

8. Secondary Outcome: Change in Fatigue Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Fatigue will be assessed at baseline and 5 weeks for each individual patient using the Patient Reported Outcomes Measurement Information System (PROMIS) Fatigue Short Form 7a v1.0 questionnaire. Raw scores are converted to standardized T scores based on national norms for patients with cancer.
  * Baseline: Mean fatigue T score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean fatigue T score for all individual patients in arm 1 (intervention)
  * Average fatigue T score for the reference population of patients with cancer is 50.0, with standard deviation of 10.0 (higher score=more fatigue)
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
T score
  Baseline | 56.79 (7.86) | 45.63 (5.53)
  week 5 timepoint: number analyzed (Participants) | 31 | 0
  week 5 timepoint | 54.51 (7.84) |

9. Secondary Outcome: Change in Sleep Disturbance Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Sleep Disturbance will be assessed at baseline and 5 weeks for each individual patient using the PROMIS Sleep Disturbance Short Form 8b v1.0 questionnaire. Raw scores are converted to standardized T scores based on national norms for patients with cancer.
  * Baseline: Mean sleep disturbance T score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean sleep disturbance T score for all individual patients in arm 1 (intervention)
  * Average sleep disturbance T score for the reference population of patients with cancer is 50.0, with standard deviation of 10.0 (higher score=more sleep disturbance)
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
T score
  Baseline | 57.44 (8.25) | 43.91 (7.99)
  week 5 timepoint: number analyzed (Participants) | 31 | 0
  week 5 timepoint | 53.85 (8.86) |

10. Secondary Outcome: Change in Physical Function Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Physical Function will be assessed at baseline and 5 weeks for each individual patient using the PROMIS Physical Function Short Form 10a v1.0 questionnaire. Raw scores are converted to standardized T scores based on national norms for patients with cancer.
  * Baseline: Mean physical function T score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean physical function T score for all individual patients in arm 1 (intervention)
  * Average physical function T score for the reference population of patients with cancer is 50.0, with standard deviation of 10.0 (higher score=better physical function)
Time Frame: 5 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T score
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
T score
  Baseline | 41.96 (5.58) | 56.60 (5.74)
  week 5 timepoint: number analyzed (Participants) | 31 | 0
  week 5 timepoint | 44.03 (6.13) |

11. Secondary Outcome: Change in Anxiety Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Anxiety will be assessed at baseline and 5 weeks for each individual patient using the Hospital Anxiety and Depression Scale.
  * Baseline: Mean anxiety score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean anxiety score for all individual patients in arm 1 (intervention)
  * Range of anxiety score 0-21 (0=no anxiety, 21=maximum anxiety)
Time Frame: 5 weeks
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 40
score on a scale
  Baseline | 6.97 (4.00) | 3.90 (2.91)
  week 4 timepoint: number analyzed (Participants) | 31 | 0
  week 4 timepoint | 5.03 (3.15) |

12. Secondary Outcome: Change in Depression Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Depression will be assessed at baseline and 5 weeks for each individual patient using the Hospital Anxiety and Depression Scale.
  * Baseline: Mean depression score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean depression score for all individual patients in arm 1 (intervention)
  * Range of depression score 0-21 (0=no depression, 21=maximum depression)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 at baseline and 1 patient in Arm 2 had missing data and the scores could not be generated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 39
score on a scale
  Baseline | 5.85 (3.38) | 1.46 (1.95)
  week 5 timepoint: number analyzed (Participants) | 31 | 0
  week 5 timepoint | 4.23 (3.96) |

13. Secondary Outcome: Change in Cognitive Difficulties - Language Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Cognitive Difficulties - Language will be assessed at baseline and 5 weeks for each individual patient using the Multiple Ability Self-Report Questionnaire.
  * Baseline: Mean language score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean language score for all individual patients in arm 1 (intervention)
  * Range of language score 0-40 (0=no language difficulties, 40=maximum language difficulties)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 at week 5 had missing data and the score could not be generated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
score on a scale
  Baseline | 15.43 (4.51) | 12.42 (3.40)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 14.83 (3.57) |

14. Secondary Outcome: Change in Cognitive Difficulties - Visual-Perceptual Ability Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Cognitive Difficulties - Visual-Perceptual Ability will be assessed at baseline and 5 weeks for each individual patient using the Multiple Ability Self-Report Questionnaire.
  * Baseline: Mean visual-perceptual ability score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean visual-perceptual ability score for all individual patients in arm 1 (intervention)
  * Range of visual-perceptual ability score 0-30 (0=no visual-perceptual difficulties, 30=maximum visual-perceptual difficulties)
Time Frame: 5 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 39
score on a scale
  Baseline | 10.79 (3.17) | 8.62 (3.39)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 10.33 (2.70) |

15. Secondary Outcome: Change in Cognitive Difficulties - Verbal Memory Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Cognitive Difficulties - Verbal Memory will be assessed at baseline and 5 weeks for each individual patient using the Multiple Ability Self-Report Questionnaire.
  * Baseline: Mean verbal memory score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean verbal memory score for all individual patients in arm 1 (intervention)
  * Range of verbal memory score 0-40 (0=no verbal memory difficulties, 40=maximum verbal memory difficulties)
Time Frame: 5 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 39
score on a scale
  Baseline | 17.15 (4.57) | 13.97 (4.36)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 16.90 (3.83) |

16. Secondary Outcome: Change in Cognitive Difficulties - Visual-Spatial Memory Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Cognitive Difficulties - Visual-Spatial Memory will be assessed at baseline and 5 weeks for each individual patient using the Multiple Ability Self-Report Questionnaire.
  * Baseline: Mean visual-spatial memory score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean visual-spatial memory score for all individual patients in arm 1 (intervention)
  * Range of visual-spatial memory score 0-40 (0=no visual-spatial memory difficulties, 40=maximum visual-spatial memory difficulties)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 at week 5 and 1 patient in Arm 2 had missing data and the scores could not be generated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 39
score on a scale
  Baseline | 14.43 (3.07) | 13.03 (4.84)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 14.53 (3.64) |

17. Secondary Outcome: Change in Cognitive Difficulties - Attention/Concentration Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Cognitive Difficulties - Attention/Concentration will be assessed at baseline and 5 weeks for each individual patient using the Multiple Ability Self-Report Questionnaire.
  * Baseline: Mean attention/concentration score for all individual patients in arm 1 (intervention)
  * 5 weeks: Mean attention/concentration score for all individual patients in arm 1 (intervention)
  * Range of attention/concentration score 0-40 (0=no attention/concentration difficulties, 40=maximum attention/concentration difficulties)
Time Frame: 5 weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 39
score on a scale
  Baseline | 17.26 (3.43) | 14.10 (3.60)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 15.83 (3.49) |

18. Secondary Outcome: Change in Objectively Assessed Pain Sensitivity Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Pain sensitivity will be assessed at baseline and 5 weeks for each individual patient using quantitative sensory testing to assess pressure pain threshold (Pain50).
  * Baseline: Mean Pain50 for all individual patients in arm 1 (intervention) and arm 2 (control)
  * 5 weeks: Mean Pain50 for all individual patients in arm 1 (intervention)
  * Range of Pain50 score: 0-10 kg/cm2 (higher number reflects higher pain threshold or lower pain sensitivity)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 had missing data at week 5 and the score could not be generated.
Measure: Mean (Standard Deviation); unit: kg/cm2
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 35 | 40
kg/cm2
  Baseline | 3.20 (1.37) | 4.06 (1.40)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 3.30 (1.38) |

19. Secondary Outcome: Change in Objectively Assessed Conditioned Pain Modulation Between Baseline and 5 Weeks of Treatment With Duloxetine
Description: Conditioned pain modulation (CPM) will be assessed at baseline and 5 weeks for each individual patient using quantitative sensory testing
  * Baseline: Mean CPM for all individual patients in arm 1 (intervention) and arm 2 (control)
  * 5 weeks: Mean CPM for all individual patients in arm 1 (intervention)
  * Range of CPM score: -60 to +60 (more positive values reflect more impaired CPM)
Time Frame: 5 weeks
Population: Only patients with pain were analyzed at week 5. Patients who discontinued study treatment early (n=4) have no data available for week 5. 1 patient in Arm 1 at baseline, 1 patient in Arm 1 at week 5, and 2 patients in Arm 2 had missing data and the scores could not be generated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
Number analyzed (Participants) | 34 | 38
score on a scale
  Baseline | 9.68 (16.47) | 7.97 (15.32)
  week 5 timepoint: number analyzed (Participants) | 30 | 0
  week 5 timepoint | 11.93 (12.76) |

ADVERSE EVENTS:
Time Frame: Adverse Event (AE) data were collected from date of study drug administration until 14 days after completion of study drug
Arm/Group | Arm 1 (Patients With Pain) | Arm 2 (Patients Without Pain -- Control)
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/40
Serious Adverse Events (participants affected / at risk) | 1/35 | 0/40
Other Adverse Events (participants affected / at risk) | 10/35 | 0/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Patients With Pain) (N=35) | Arm 2 (Patients Without Pain -- Control) (N=40)
congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1 (Patients With Pain) (N=35) | Arm 2 (Patients Without Pain -- Control) (N=40)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 0 (0)
insomnia (Psychiatric disorders) | 3 (3) | 0 (0)
fatigue (General disorders) | 2 (2) | 0 (0)
nausea (Gastrointestinal disorders) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/12/NCT01912612/Prot_SAP_000.pdf